CLINICAL TRIAL: NCT03790319
Title: Scientific Evaluation of Trainings for Emotional Competence, Compassion and Relationship Competences
Brief Title: Emotional Competence and Compassion Training
Acronym: ECCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ECCT
Record Dates: First submitted 2018-12-14; First posted 2018-12-31 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Emotional Intelligence
Keywords: Stress; Emotion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single Workshop 'The Emotional Backpack': Subjects of this group are participating in one single workshop over three days.
  Interventions: Behavioral: The Emotional Backpack
- Year Program 'The Power of Feelings': Subjects of this group are participating in three workshops of over 3 days each in a continuing group over nine months. They are animated to deal with the content inbetween the workshops through biweekly e-mails and to exchange in couples.
  Interventions: Behavioral: The Power of Feelings

INTERVENTIONS:
Behavioral: The Power of Feelings — Three workshops of three days each teach about the five basic feelings rage, sadness, fear, shame and joy and talk about the powerful and destructive qualities they can have. In addition to that they are about how to deal with emotions, which are defined as unfelt feelings of the past.
  Smaller lectures give the participants an overview about the themes. Through exercises the participants can make experiences p.e. about each of the feelings. Another element is the sharing in dyads or small groups about actual feelings to practice emotional disclosure and to build a culture of openness and compassion.
  Groups: Year Program 'The Power of Feelings'
Behavioral: The Emotional Backpack — One workshop of three days teach about how to deal with emotions, which are defined as unfelt feelings of the past. They show a way to work in couples with a form of emotional disclosure that helps process emotions that have been overwhelming in the past.
  Smaller lectures give the participants an overview about the themes. Through exercises the participants can make experiences p.e. about each of the feelings. Another element is the sharing in dyads or small groups about actual feelings to practice emotional disclosure and to build a culture of openness and compassion.
  Groups: Single Workshop 'The Emotional Backpack'

SUMMARY:
In this study several different face-to-face workshops about emotional competence and compassion are scientifically evaluated with psychometric questionnaires and heart rate variability measuring.

DETAILED DESCRIPTION:
Stress and stress related diseases are a huge health burden in modern societies. Psycho-emotional stress plays a key role in stress regulation. Therefore this study aims to investigate the effects of online-courses addressing emotion regulation.

For this aim several different workshops about emotional competence and compassion are scientifically evaluated with psychometric questionnaires and heart rate variability measuring. The workshops are planned by the trainers and people register on their own initiative.

The seminars are either single workshops over three days or a yearly program consisting of three three-day-workshops. They consist of lectures and exercises about the character of the different feelings, about the characteristics of emotions and teach practices on how to dael with difficult emotions.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years
* participation in one of the included courses
* e-mail address

Exclusion Criteria:

* participation in another study
* no verbal communication (german) possible
* dementia or another disease that limits cognitive abilities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults who enrolled themselves from their own initiative into one of the included courses
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-Report Measure for the Assessment of Emotion Regulation Skills (SEK-27) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-108, higher score meaning a better outcome

SECONDARY OUTCOMES:
The Saarbrücken Personality Questionnaire (SPF) based on the Interpersonal Reactivity Index (IRI) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 16-80, higher score meaning a better outcome
The World Health Organisation- Five Well-Being Index (WHO-5) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  assessing full scale, range 0-100, higher score meaning a better outcome
General Self-efficacy Short Scale (ASKU) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 3-15, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-42, lower score meaning a better outcome
Mindful Attention Awareness Scale (MAAS) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 15-90, higher score meaning a better outcome
Perceived Stress Scale (PSS-10) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-40, lower score meaning a better outcome
Medical Outcomes Study Short Form (MOS SF-36) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-100, higher score meaning a better outcome
Heart Rate Variability (HRV) | Assessing change from baseline to 3 and 6 months after baseline in the yearly program
  24h measuring

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Charité Medical University, Department of Integrative Medicine at the Immanual Hospital Berlin, Berlin, Germany